CLINICAL TRIAL: NCT00061295
Title: Body Weight Supported Ambulation Training After Spinal Cord Injury
Brief Title: Treadmill Training With Body Weight Support in Patients With Spinal Cord Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01HD037460-01 (NIH)
Record Dates: First submitted 2003-05-23; First posted 2003-05-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: Spinal Cord Injury
Keywords: Locomotion; Spinal Cord Injury; Body Weight Supported Walking
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Body weight support treadmill training

SUMMARY:
Body weight support (BWS) treadmill training uses an overhead harness to give partial support to patients walking on a treadmill. This study will determine whether BWS training is more effective than conventional rehabilitation therapy in improving walking ability in patients with spinal cord injuries (SCI).

DETAILED DESCRIPTION:
Gait rehabilitation is a specific component of physical rehabilitation of persons with sub-acute or chronic spinal cord injury (SCI). One novel method of gait rehabilitation involves the use of an overhead support point and a harness. The BWS strategy has been combined with treadmill-based gait training in recent studies with dramatic results. It is believed that this form of training may enhance output of a 'central pattern generator' of stepping movement from circuitry intrinsic to the patient's spinal cord. However, only limited attention has been paid to the role that training-induced physical conditioning might play in mediating functional improvements.

This study will evaluate whether BWS gait training is more effective than conventional rehabilitation therapy in improving functional gait in patients with neurologically incomplete spinal cord injury. The study will also compare treadmill-based training to overground-based training. Treadmill-based training has the inherent advantage of providing highly rhythmic input to the subject's legs; overground-based training has the inherent advantage of allowing use of assistive devices and thereby replicating a more 'natural' training condition.

Patients with chronic SCI (greater than 1 year post-injury) and patients with sub-acute SCI (2 to 8 months post-injury) will be evaluated. Patients with chronic SCI will be randomly assigned to one of 3 groups: body weight support and treadmill-based training, body weight support and overground training, and conventional rehabilitation therapy. Patients with sub-acute injury will be randomized to receive either BWS treadmill training or conventional rehabilitation. Training sessions are typically 1 hour long, with 3 sessions per week for 13 weeks.

All patients will be evaluated with a battery of functional, metabolic, and neurophysiologic measures prior to the onset of training and during the week after training has been completed. The primary outcome measure will be average maximum overground walking velocity without body weight support but with the use of passive assistive devices. Secondary measures will concentrate on function (balance, mobility), fitness (work capacity, strength, gait efficiency), and spinal cord neurophysiology (motor conduction, reflex excitability).

ELIGIBILITY:
Inclusion Criteria for Patients with Chronic Injury:

* Spinal cord injury at or above the T10 spine
* 1 year post injury
* Some volitional movement in one or both limbs (i.e., motor incomplete)
* Ability to stand with limited bracing
* Ability to rise from sit to stand with no more that moderate assistance

Inclusion Criteria for Patients with Subacute Injury:

* Spinal cord injury at or above the T10 spine
* 2 to 8 months post injury
* Volitional movement in at least one lower limb muscle (i.e., motor incomplete), although may not be capable of unsupported standing or moving from sit-to-stand without maximal assistance

Exclusion Criteria:

* Fractures at or below T11
* Neoplastic, degenerative, or vascular disorders of the spine or spinal cord
* Significant orthopaedic conditions that would interfere with regular exercise or rehabilitation therapy
* Decubitus ulcer
* Advanced urinary tract infection
* Medical conditions that increase the probability of having a seizure in response to single pulse transcranial magnetic stimulation

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-03; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Blair M. Calancie, Principal Investigator — University of Miami Project to Cure Paralysis
Locations (1):
- Upstate Medical University, Miami, Florida, United States